CLINICAL TRIAL: NCT07314229
Title: Prevalence of Exercise-induced Ventilatory Limitation and Associated Factors in Patients With Cystic Fibrosis Receiving Elexacaftor-Tezacaftor-Ivacaftor
Acronym: MUCOLIMEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024_0277; 2024-A02709-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-11-24; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis (CF); Mucoviscidosis
Keywords: Cystic fibrosis; physical activity; CFTR modulator treatment; exercise limitation; respiratory physiology; ventilatory limitation; reduction in ventilatory reserve; dynamic distension
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: No control group. Patients treated with ETI (Kaftrio-Kalydeco©) are treated as part of the management of their condition in accordance with the indications for marketing authorisation (MA), temporary authorisation for use (ATU) or French compassionate access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients treated with ETI (Kaftrio-Kalydeco©) (Experimental)
  Interventions: Device: Measurement of resistance through forced oscillations and continuous measurement of ventilation and inspiratory capacity during TM6

INTERVENTIONS:
Device: Measurement of resistance through forced oscillations and continuous measurement of ventilation and inspiratory capacity during TM6 — Measurement of resistance through forced oscillations and continuous measurement of ventilation and inspiratory capacity during TM6

SUMMARY:
Cystic fibrosis is a genetic disorder affecting the entire body and associated with respiratory exacerbations, impaired quality of life and reduced life expectancy. The therapeutic management of cystic fibrosis has been profoundly changed by the recent arrival of a combination of highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators, Elexacaftor-Tezacaftor-Ivacaftor (ETI), which improve quality of life, respiratory function and reducing the number of exacerbations. The impact of these treatments on exercise adaptation has not been clearly identified.

The main objective is to estimate the prevalence of ventilatory reserve amputation during submaximal exercise testing assessed by the 6-minute walk test (6MWT) in patients with cystic fibrosis treated with ETIs.

DETAILED DESCRIPTION:
Cystic fibrosis is a genetic disorder affecting the entire body and associated with respiratory exacerbations, impaired quality of life and reduced life expectancy. The therapeutic management of cystic fibrosis has been profoundly changed by the recent arrival of a combination of highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators, Elexacaftor-Tezacaftor-Ivacaftor (ETI), which improve quality of life, respiratory function and reducing the number of exacerbations. The impact of these treatments on exercise adaptation has not been clearly identified.

The main objective is to estimate the prevalence of ventilatory reserve amputation during submaximal exercise testing assessed by the 6-minute walk test (6MWT) in patients with cystic fibrosis treated with ETIs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult aged 18 or over
* Suffering from cystic fibrosis
* Treated at the CRCM in Lille and Créteil
* Treated by ETI
* Be covered by social security
* Be able to understand the requirements of the study, provide written informed consent, and comply with the study's data collection procedures

Exclusion Criteria:

* Medical contraindication or inability to perform a stress test according to ERS recommendations

  * Absolute contraindications
  * Relative contraindications:
* Exacerbation of the condition in the 4 weeks preceding the V1 visit (27).
* Pregnant or breastfeeding women
* Administrative reasons
* Persons deprived of their liberty
* Minors or protected adults
* Persons who have refused or are unable to give informed consent
* Persons in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of ventilatory limitation measured by a portable spirometer during a submaximal exercise test (6-minute walk test) in patients with cystic fibrosis undergoing ETI. | duration of 56 weeks starting in December 2025
  The primary endpoint is ventilatory limitation defined as the difference between the estimated theoretical maximun minute ventilatory volume (VMM in L/min) estimated by multiplying FEV1 (L) x 35 and the measurement of external ventilation during exercise (VE, L/min) using a portable spirometer divided by the theoretical VM x100 less than 15%.
  Ventilatory limitation = (MMV (L/min) - VE (L/min) /MMV (L/min))*100 < 15%

SECONDARY OUTCOMES:
Estimate the prevalence of ventilatory limitation measured using a portable spirometer during a maximal incremental step test (A-STEP) with progressive steps in patients with cystic fibrosis undergoing ETI. | duration of 56 weeks starting in December 2025
  The assessment criterion is the difference between the estimated theoretical maximun minute ventilatory volume (VMM in L/min) estimated by multiplying FEV1 (L) x 35 and the measurement of external ventilation (VE in L/min) using a portable spirometer during exercise divided by the theoretical VM x100 less than 15%.
Assessment of the prevalence of dynamic distension during a submaximal (TM6) or maximal (incremental step test according to the A-Step protocol) exercise test by spirometry | duration of 56 weeks starting in December 2025
  The criterion for judgement is a decrease in inspiratory capacity (L) of more than 150 mL within 30 seconds after the end of the effort compared to the pre-effort inspiratory capacity (L) measured by spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided